CLINICAL TRIAL: NCT00442585
Title: Double Blind, Randomised, Parallel Group, Placebo Controlled Clinical Trial of S(+)-Ibuprofen Effects on TxB2 Concentrations and Platelet Aggregation in Aspirin-treated Healthy Adult Volunteers
Brief Title: S(+)-Ibuprofen Effects on Asprin Treated Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gebro Pharma GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gebro-I-24-13; EUDRACT 2006-002159-33
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S(+)-ibuprofen

SUMMARY:
The purpose of this clinical trial is to determine whether S(+)-ibuprofen affect the platelet inhibition under steady state acetylsalicylic acid conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian volunteer
* Must be able to swallow tablets

Exclusion Criteria:

* Underlying diseases
* Ulcus pepticum in history
* Abuse of alcoholic beverages (40g/d)
* Hypersensitivity to investigational medicinal products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72
Dates: Start 2006-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage of inhibition of TxB2 after 1, 3, 7 and 10 days

SECONDARY OUTCOMES:
percentage of subjects with >90% inhibition of TxB2, CEPI-CT and CADP-CT measured by PAF100,
prostacyclin metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Christian Joukhadar, MD, Principal Investigator — Department of Clinical Pharmacology, Division of Clinical Pharmacokinetics, Medical Univerisity of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Cryer B, Berlin RG, Cooper SA, Hsu C, Wason S. Double-blind, randomized, parallel, placebo-controlled study of ibuprofen effects on thromboxane B2 concentrations in aspirin-treated healthy adult volunteers. Clin Ther. 2005 Feb;27(2):185-91. doi: 10.1016/j.clinthera.2005.01.011. PMID 15811481